CLINICAL TRIAL: NCT06361433
Title: Phase I/II Trial of Intracerebral Transplantation of Autologous Bone Marrow Stromal Cells Combined With Recombinant Peptide Scaffold for Patients With Chronic Intracerebral Hemorrhage
Brief Title: Intracerebral Transplantation of Autologous MSC Combined With Scaffold Product for Chronic Intracerebral Hemorrhage
Acronym: RAINBOW-Hx
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hokkaido University Hospital (Other)
Collaborators: Japan Agency for Medical Research and Development (Other Government)
Responsible Party: Principal Investigator, Masahito Kawabori, Lecturer, Hokkaido University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R5-11
Record Dates: First submitted 2024-01-25; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Intracerebral Hemorrhage
Keywords: Mesenchymal stromal cell; scaffold; chronic; intracerebral hemorrhage; intraparenchymal transplantation
MeSH Terms: conditions — Cerebral Hemorrhage; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cell product transplantation (Experimental): Autologous MSC with scaffold containing approximately 5 x 10^7 MSC cells.
  Interventions: Drug: HUFF-01

INTERVENTIONS:
Drug: HUFF-01 — autologous MSC combined with scaffold

SUMMARY:
The goal of this clinical trial is to test intracerebral transplantation of stem cell product in patient with chronic intracerebral hemorrhage. The main questions aims to answer are:

* The safety of the product
* The efficacy of the product

DETAILED DESCRIPTION:
Introduction:

Intracerebral hemorrhage stands as a leading global cause of death and disability, posing a significant challenge with limited treatment options, especially for chronic patients. Recent advances of stem cell therapies have opened new avenues for therapeutic potential. The investigators' previous preclinical research has demonstrated that intracerebral transplantation of bone marrow stromal cells (BMSCs) combined with a recombinant human collagen type I scaffold enables higher cell survival and engraftment, holds promising potential. The investigators present the protocol for a novel clinical trial, named "Research on Advanced Intervention using Novel Bone Marrow Stem Cells for Chronic Intracerebral Hemorrhage" (RAINBOW-Hx).

Methods and Analysis:

RAINBOW-Hx is a phase I/II, open-label, uncontrolled study with the primary objective of assessing the safety and efficacy of intracerebral transplantation of autologous BMSCs combined with the scaffold (HUFF-01) in patients with chronic intracerebral hemorrhage. Eight patients, experiencing moderate to severe neurological deficits for 12 months or longer, will be enrolled. The hemorrhage location will be limited to the basal ganglia and thalamus. Approximately 50 mL of bone marrow will be extracted from the iliac bone of each patient, and BMSCs will be cultured using autologous platelet lysate. Three days before transplantation, BMSCs will be combined with the scaffold to generate HUFF-01. Each patient will receive a 50,000 HUFF-01 dose, containing approximately 50 million BMSCs, through stereotactic transplantation into the hemorrhagic cavity. Neurological assessments, magnetic resonance imaging, 18F-fluorodeoxyglucose positron emission tomography, and 123I-Iomazenil single-photon emission computed tomography will be performed for one year after administration.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 20 and 70 years
* 2. Clinical diagnosis of intracerebral hemorrhage 12 month or more from onset
* 3. Hemorrhagic location of unilateral basal ganglia or thalamus
* 4. Moderate to severe neurological symptoms; mRS 3 or 4, and Brunnstrom stage Ⅲ or IV
* 5. No significant neurological impairment before hemorrhage (Pre-hemorrhagic mRS of 0 or 1)
* 6. Subjects who can give informed consent by its self

Exclusion Criteria:

* 1. Severe microbleeds found by T2*
* 2. Hemorrhagic cavity less than 2 mL
* 3. The hemorrhage is due to arteriovenous malformation, cerebral aneurysm, and Moyamoya disease
* 4. Subject showing obvious communication between the hemorrhagic cavity and lateral ventricle on MRI
* 5. Subject showing severe lower extremity contracture (Maximum knee extension less than -15 degrees, Maximum ankle flexion less than 0 degree)
* 6. Subject's body weight less than 45 kg for male and 40kg for female
* 7. Anaemia (Hg < 10·0 g/dL)
* 8. Thrombocytopaenia (platelet count < 100,000/mm3)
* 9. Severe heart disease (ischaemic heart disease, heart failure)
* 10. Uncontrolled hypertension, despite antihypertensive therapy
* 11. Carriers of infectious disease: syphilis, HBV, HCV, HIV-1/HIV-2, HTLV-1, parvovirus B19
* 12. Pregnant or lactating or expecting to become pregnant during the study
* 13. History of malignancy
* 14. Systemic organ failure ALT ≤ 3·0× upper limit of normal Total bilirubin ≤ 1·5× upper limit of normal Serum creatinine ≤ 1·5× upper limit of normal
* 15. Known serious allergy to any agents used in the study
* 16. Contraindication for magnetic resonance imaging
* 17. Any condition that in the judgement of the investigator would place the patient at undue risk

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | one year
  Listing unexpected CTCAE grade changes in physiological (physical examination/blood test) and Radiographical (MRI/CT) examination

SECONDARY OUTCOMES:
Change in mRS examination | One year
  Percentage of the patients number who showed improvement of mRS (0-6, higher score means worse outcome) of more than 1 point
Change in NIHSS examination | One year
  Mean improvement of NIHSS (0-42, higher score means worse outcome)
Change in FIM examination | One year
  Mean improvement of FIM (18-126, higher score means better outcome)
Change in Fugl-Myer examination | One year
  Mean improvement of Fugl-Myer (0-226, higher score means better outcome)
Change in Barthal index examination | One year
  Mean improvement of Barthal index (0-100, higher score means better outcome)
Change in FDG-PET examination | One year
  Mean improvement of FDG-PET set for ipsilateral motor cortex
Change in IMZ-SPECT examination | One year
  Mean improvement of IMZ-SPECT set for ipsilateral motor cortex

CONTACTS AND LOCATIONS:
Locations (1):
- Hokkaido University Hospital, Sapporo, Hokkaido, Japan

IPD SHARING:
Plan to Share IPD: No